CLINICAL TRIAL: NCT01141478
Title: Randomized Controlled Trial of Proton Beam Radiotherapy + Sorafenib vs. Sorafenib for Patients With Hepatocellular Carcinoma Exceeding San Francisco Criteria
Brief Title: Proton Radiotherapy Plus Sorafenib Versus Sorafenib for Patients With HCC Exceeding San Francisco Criteria
Acronym: HCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to low enrollment
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5100104
Record Dates: First submitted 2010-05-24; First posted 2010-06-10 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; Proton Beam Radiotherapy; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Proton Beam Radiotherapy plus Sorafenib (Active Comparator): A combination of radiation therapy (proton) to kill tumor cells as well as Sorafenib which is a study drug administered to patients to stop tumor growth.
  Interventions: Radiation: Proton Beam Radiotherapy; Drug: Sorafenib
- Sorafenib (Active Comparator): Sorafenib is an oral pill taken daily to inhibit tumor growth at the cellular level.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Radiation: Proton Beam Radiotherapy — Fifteen consecutive sessions
  Arms: Proton Beam Radiotherapy plus Sorafenib
Drug: Sorafenib — 400 mg po bid

SUMMARY:
This study is designed to determine whether proton beam radiotherapy plus Sorafenib compared to Sorafenib alone will produce the best results for treating patients with Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are candidates to receive both proton beam and sorafenib
2. Patients with tumor burden that exceeds San Francisco criteria

Exclusion Criteria:

1. Patients who are candidates for surgical resection
2. Patients with tumor burden within Milan and/or San Francisco criteria
3. Patients who have contraindication to receive proton
4. Patients with contraindication to receive sorafenib including uncontrolled hypertension, coumadin treatment and prior intolerability to the drug
5. Patients treated previously by any locoregional treatment
6. Patients with prior liver transplant
7. Patients with child class C
8. Patients with model for end-stage liver disease (MELD) score of > 25
9. Patients with other comorbid diseases that may impact survival
10. Patients with ongoing alcohol intake
11. Patients with active sepsis
12. Patients with gastrointestinal bleeding within a week
13. Patients unwilling to sign informed consent form
14. Patients with history of noncompliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09-08 (Actual); Primary Completion 2014-12-26 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael deVera, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Beam Radiotherapy Plus Sorafenib | Sorafenib
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proton Beam Radiotherapy Plus Sorafenib | Sorafenib | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
Alfa-feto protein [Mean (Standard Deviation); unit: ng/ml] — Reference range for 0 - 100 years -All 0 - 8.7 ng/ml Baseline alpha feto protein levels were measured not to serve as a measure of eligibility or outcomes, but simply as another marker for the diagnosis of hepatocellular carcinoma. Population: 8 subjects were consented. 4 to Arm A, and 4 to Arm B. However, 2 subjects (one from each arm) withdrew consent or were lost to follow up leaving 6 subjects total to be analyzed.
  ng/ml
    number analyzed (Participants) | 3 | 3 | 6
    (all) | 1413.8 (1777) | 44319 (29640.2) | 22866.4 (30082.1)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate Between Time of Consent and Time of Death
Description: All subjects are to be followed from time of consent until time of death. Subjects in both arms will require either a CT scan or MRI of the abdomen every three months to monitor tumor progression. Follow up imaging with be the same modality used at baseline (CT or MRI). All subjects are to be evaluated in the liver clinic 4 weeks after treatment and then every 3 months. Subjects in the Proton arm will require a CT or MRI 4-6 weeks after treatment and then every three months. Subjects receiving Proton therapy will also be followed in the radiation medicine clinic by their treating radiation oncologist every 3 months for the first year and then every 6 months.
Time Frame: Change between time of informed consent and primary completion date of study, an average of 4 years per participant
Population: two subjects withdrew prior to over all survival rate measurement
Measure: Mean (Full Range); unit: years
Arm/Group | Proton Beam Radiotherapy Plus Sorafenib | Sorafenib
Number analyzed (Participants) | 3 | 3
years | 1.6 [0.1 to 3.7] | 0.36 [0.3 to 0.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment to death or time when a patient was lost to follow-up
Description: All subjects are at risk for serious and non serious adverse events due to the progression of their liver disease and the possible side effects from both study treatment arms.
Arm/Group | Proton Beam Radiotherapy Plus Sorafenib | Sorafenib
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Radiotherapy Plus Sorafenib (N=4) | Sorafenib (N=4)
Death - cerebral hemorrahic stroke (General disorders) | 1 (1) | 0 (0) — Subject randomized to Arm "A" - received 5 proton treatments starting 11/2010 to 12/2010, had a cerebral hemorrhage 5/2014 and expired. This incident was rated as possibly related to treatment yet expected in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No